CLINICAL TRIAL: NCT03548935
Title: Effect and Safety of Semaglutide 2.4 mg Once-weekly in Subjects With Overweight or Obesity
Brief Title: STEP 1: Research Study Investigating How Well Semaglutide Works in People Suffering From Overweight or Obesity
Acronym: STEP 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9536-4373; U1111-1200-8053 (Other: World Health Organization (WHO)); 2017-003436-36 (Registry Identifier: European Medicines Agency (EudraCT))
Record Dates: First submitted 2018-05-25; First posted 2018-06-07 (Actual); Results first posted 2021-08-11 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Metabolism and Nutrition Disorder; Overweight or Obesity
MeSH Terms: conditions — Nutrition Disorders; Overweight; Obesity | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Semaglutide s.c. 2.4 mg once weekly (Experimental): Participants will receive semaglutide for 68 weeks.
  Interventions: Drug: Semaglutide
- Semaglutide placebo (Placebo Comparator): Participants will receive semaglutide matching placebo for 68 weeks.
  Interventions: Drug: Placebo (semaglutide)

INTERVENTIONS:
Drug: Semaglutide — Participants will receive semaglutide subcutaneous (s.c.; under the skin) injection(s) once-weekly as well as diet and physical activity counselling for 68 weeks. Dose escalation of semaglutide will take place as follows: 0.25 mg from week 1 to 4, 0.5 mg from week 5 to 8, 1.0 mg from week 9 to 12, 1.7 mg from week 13 to 16 and 2.4 mg from week 17 to week 68.
  Arms: Semaglutide s.c. 2.4 mg once weekly
Drug: Placebo (semaglutide) — Participants will receive semaglutide matching placebo s.c. injection(s) once-weekly as well as diet and physical activity counselling for 68 weeks.
  Arms: Semaglutide placebo

SUMMARY:
This study will look at the change in participants' body weight from the start to the end of the study. The weight loss in participants taking semaglutide (a new medicine) will be compared to the weight loss of participants taking "dummy" medicine. In addition to taking the medicine, participants will have talks with study staff about healthy food choices, how to be more physically active and what you can do to lose weight. Participants will either get semaglutide or "dummy" medicine - which treatment participants get, is decided by chance. Participants will need to take 1 injection once a week. The study medicine is injected with a thin needle in a skin fold in the stomach, thigh or upper arm. The study has two phases: A main phase and an extension phase.The main phase will last for about 1.5 years. Participants will have 15 clinic visits and 10 phone calls with the study doctor. Extension phase: Approximately 300 participants will continue in the extension phase in the following countries only: Canada, Germany, the UK and selected sites in the US and Japan. These participants will be in the study for about 2.5 years.They will not receive treatment, but will attend another 5 follow-up visits with the study doctor.

ELIGIBILITY:
Inclusion Criteria:

Main phase:

* Male or female, age greater than or equal to 18 years at the time of signing informed consent
* Body mass index (BMI) greater than or equal to 30.0 kg/sqm or greater than or equal to 27.0 kg/sqm with the presence of at least one of the following weight-related comorbidities (treated or untreated): hypertension, dyslipidaemia, obstructive sleep apnoea or cardiovascular disease
* History of at least one self-reported unsuccessful dietary effort to lose body weight

Extension phase:

* Informed consent for the extension phase obtained before any trial related activities for the extension phase
* On randomised treatment on the target dose at week 68, i.e. treated with 2.4 mg semaglutide once-weekly or semaglutide placebo

Exclusion Criteria:

Main phase:

* Glycated haemoglobin (HbA1C) greater than or equal to 48 mmol/mol (6.5%) as measured by the central laboratory at screening
* A self-reported change in body weight greater than 5 kg (11 lbs) within 90 days before screening irrespective of medical records

Extension phase:

* Female who is pregnant or intends to become pregnant during the extension phase
* Any disorder, unwillingness or inability, not covered by any of the other exclusion criteria, which in the investigator's opinion, might jeopardise the subject's compliance with the extension of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1961 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2021-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (114):
- United States (35):
  - Novo Nordisk Investigational Site, Anniston, Alabama
  - Novo Nordisk Investigational Site, Anaheim, California
  - Novo Nordisk Investigational Site, Lomita, California
  - Novo Nordisk Investigational Site, Spring Valley, California
  - Novo Nordisk Investigational Site, Aurora, Colorado
  - Novo Nordisk Investigational Site, Waterbury, Connecticut
  - Novo Nordisk Investigational Site, Chiefland, Florida
  - Novo Nordisk Investigational Site, Crystal River, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Ocala, Florida
  - Novo Nordisk Investigational Site, Panama City, Florida
  - Novo Nordisk Investigational Site, Plantation, Florida
  - Novo Nordisk Investigational Site, Ponte Vedra, Florida
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Topeka, Kansas
  - Novo Nordisk Investigational Site, Louisville, Kentucky
  - Novo Nordisk Investigational Site, Buckley, Michigan
  - Novo Nordisk Investigational Site, City of Saint Peters, Missouri
  - Novo Nordisk Investigational Site, Butte, Montana
  - Novo Nordisk Investigational Site, Omaha, Nebraska
  - Novo Nordisk Investigational Site, Rochester, New York
  - Novo Nordisk Investigational Site, Salisbury, North Carolina
  - Novo Nordisk Investigational Site, Wilmington, North Carolina
  - Novo Nordisk Investigational Site, West Reading, Pennsylvania
  - Novo Nordisk Investigational Site, Charleston, South Carolina
  - Novo Nordisk Investigational Site, Simpsonville, South Carolina
  - Novo Nordisk Investigational Site, Nashville, Tennessee
  - Novo Nordisk Investigational Site, Austin, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Round Rock, Texas
  - Novo Nordisk Investigational Site, Bountiful, Utah
  - Novo Nordisk Investigational Site, Richmond, Virginia
  - Novo Nordisk Investigational Site, Renton, Washington
- Argentina (5):
  - Novo Nordisk Investigational Site, CABA
  - Novo Nordisk Investigational Site, Ciudad de Buenos Aires
  - Novo Nordisk Investigational Site, Corrientes
  - Novo Nordisk Investigational Site, Córdoba
  - Novo Nordisk Investigational Site, Santa Rosa
- Belgium (5):
  - Novo Nordisk Investigational Site, Boussu
  - Novo Nordisk Investigational Site, Brussels
  - Novo Nordisk Investigational Site, Edegem
  - Novo Nordisk Investigational Site, Leuven
  - Novo Nordisk Investigational Site, Liège
- Bulgaria (2):
  - Novo Nordisk Investigational Site, Plovdiv
  - Novo Nordisk Investigational Site, Sofia
- Canada (6):
  - Novo Nordisk Investigational Site, Edmonton, Alberta
  - Novo Nordisk Investigational Site, Surrey, British Columbia
  - Novo Nordisk Investigational Site, Hamilton, Ontario
  - Novo Nordisk Investigational Site, North York, Ontario
  - Novo Nordisk Investigational Site, Toronto, Ontario
  - Novo Nordisk Investigational Site, Québec
- Novo Nordisk Investigational Site, Aarhus N, Denmark
- Finland (2):
  - Novo Nordisk Investigational Site, Oulu
  - Novo Nordisk Investigational Site, University of Helsinki
- France (6):
  - Novo Nordisk Investigational Site, Le Coudray
  - Novo Nordisk Investigational Site, Narbonne
  - Novo Nordisk Investigational Site, Paris
  - Novo Nordisk Investigational Site, Pessac
  - Novo Nordisk Investigational Site, Pierre-Bénite
  - Novo Nordisk Investigational Site, Vénissieux
- Germany (12):
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Bochum
  - Novo Nordisk Investigational Site, Essen
  - Novo Nordisk Investigational Site, Falkensee
  - Novo Nordisk Investigational Site, Frankfurt
  - Novo Nordisk Investigational Site, Giessen
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Hohenmölsen
  - Novo Nordisk Investigational Site, Leipzig
  - Novo Nordisk Investigational Site, Saint Ingbert-Oberwürzbach
  - Novo Nordisk Investigational Site, Stuttgart
  - Novo Nordisk Investigational Site, Wangen
- India (12):
  - Novo Nordisk Investigational Site, Guntur, Andhra Pradesh
  - Novo Nordisk Investigational Site, Secunderabad,, Andhra Pradesh
  - Novo Nordisk Investigational Site, Surat, Gujarat
  - Novo Nordisk Investigational Site, Rohtak, Haryana
  - Novo Nordisk Investigational Site, Thiruvananthapuram, Kerala
  - Novo Nordisk Investigational Site, Nagpur, Maharashtra
  - Novo Nordisk Investigational Site, Pune, Maharashtra
  - Novo Nordisk Investigational Site, New Dehli, New Delhi
  - Novo Nordisk Investigational Site, Chennai, Tamil Nadu
  - Novo Nordisk Investigational Site, Kolkata, West Bengal
  - Novo Nordisk Investigational Site, Hyderabad
  - Novo Nordisk Investigational Site, Ludhiana
- Japan (3):
  - Novo Nordisk Investigational Site, Chiba-shi, Chiba
  - Novo Nordisk Investigational Site, Suita-shi, Osaka
  - Novo Nordisk Investigational Site, Tokyo
- Mexico (3):
  - Novo Nordisk Investigational Site, Guadalajara, Jalisco
  - Novo Nordisk Investigational Site, Hermosillo, Sonora
  - Novo Nordisk Investigational Site, Mérida, Yucatán
- Poland (4):
  - Novo Nordisk Investigational Site, Gdynia
  - Novo Nordisk Investigational Site, Lodz
  - Novo Nordisk Investigational Site, Poznan
  - Novo Nordisk Investigational Site, Szczecin
- Novo Nordisk Investigational Site, San Juan, Puerto Rico
- Russia (7):
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Novosibirsk
  - Novo Nordisk Investigational Site, Penza
  - Novo Nordisk Investigational Site, Saint Petersburg
  - Novo Nordisk Investigational Site, Tomsk
  - Novo Nordisk Investigational Site, Voronezh
  - Novo Nordisk Investigational Site, Yaroslavl
- Novo Nordisk Investigational Site, Taipei, Taiwan
- United Kingdom (9):
  - Novo Nordisk Investigational Site, Bristol
  - Novo Nordisk Investigational Site, Cambridge
  - Novo Nordisk Investigational Site, Coventry
  - Novo Nordisk Investigational Site, Glasgow
  - Novo Nordisk Investigational Site, Liverpool
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Norwich
  - Novo Nordisk Investigational Site, Rotherham
  - Novo Nordisk Investigational Site, Taunton

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com/sharing-results

REFERENCES:
- [Background] Kushner RF, Calanna S, Davies M, Dicker D, Garvey WT, Goldman B, Lingvay I, Thomsen M, Wadden TA, Wharton S, Wilding JPH, Rubino D. Semaglutide 2.4 mg for the Treatment of Obesity: Key Elements of the STEP Trials 1 to 5. Obesity (Silver Spring). 2020 Jun;28(6):1050-1061. doi: 10.1002/oby.22794. PMID 32441473
- [Result] Wilding JPH, Batterham RL, Calanna S, Davies M, Van Gaal LF, Lingvay I, McGowan BM, Rosenstock J, Tran MTD, Wadden TA, Wharton S, Yokote K, Zeuthen N, Kushner RF; STEP 1 Study Group. Once-Weekly Semaglutide in Adults with Overweight or Obesity. N Engl J Med. 2021 Mar 18;384(11):989-1002. doi: 10.1056/NEJMoa2032183. Epub 2021 Feb 10. PMID 33567185
- [Derived] Schattenberg JM, Gronbaek H, Kliers I, Ladelund S, Long MT, Nygard SB, Sanyal AJ, Davies MJ. Proteomic signatures reflect effects of semaglutide treatment for MASH. JHEP Rep. 2025 Jul 22;7(10):101521. doi: 10.1016/j.jhepr.2025.101521. eCollection 2025 Oct. PMID 40980163
- [Derived] Kral P, Holst-Hansen T, Olivieri AV, Ivanescu C, Lamotte M, Larsen S. The Correlation Between Body Mass Index and Health-Related Quality of Life: Data from Two Weight Loss Intervention Studies. Adv Ther. 2024 Nov;41(11):4228-4247. doi: 10.1007/s12325-024-02932-8. Epub 2024 Sep 24. PMID 39316288
- [Derived] Wadden TA, Brown GK, Egebjerg C, Frenkel O, Goldman B, Kushner RF, McGowan B, Overvad M, Fink-Jensen A. Psychiatric Safety of Semaglutide for Weight Management in People Without Known Major Psychopathology: Post Hoc Analysis of the STEP 1, 2, 3, and 5 Trials. JAMA Intern Med. 2024 Nov 1;184(11):1290-1300. doi: 10.1001/jamainternmed.2024.4346. PMID 39226070
- [Derived] McGowan BM, Houshmand-Oeregaard A, Laursen PN, Zeuthen N, Baker-Knight J. Impact of BMI and comorbidities on efficacy of once-weekly semaglutide: Post hoc analyses of the STEP 1 randomized trial. Obesity (Silver Spring). 2023 Apr;31(4):990-999. doi: 10.1002/oby.23732. Epub 2023 Mar 6. PMID 36876594
- [Derived] Heerspink HJL, Apperloo E, Davies M, Dicker D, Kandler K, Rosenstock J, Sorrig R, Lawson J, Zeuthen N, Cherney D. Effects of Semaglutide on Albuminuria and Kidney Function in People With Overweight or Obesity With or Without Type 2 Diabetes: Exploratory Analysis From the STEP 1, 2, and 3 Trials. Diabetes Care. 2023 Apr 1;46(4):801-810. doi: 10.2337/dc22-1889. PMID 36801984
- [Derived] Kosiborod MN, Bhatta M, Davies M, Deanfield JE, Garvey WT, Khalid U, Kushner R, Rubino DM, Zeuthen N, Verma S. Semaglutide improves cardiometabolic risk factors in adults with overweight or obesity: STEP 1 and 4 exploratory analyses. Diabetes Obes Metab. 2023 Feb;25(2):468-478. doi: 10.1111/dom.14890. Epub 2022 Oct 28. PMID 36200477
- [Derived] Perreault L, Davies M, Frias JP, Laursen PN, Lingvay I, Machineni S, Varbo A, Wilding JPH, Wallenstein SOR, le Roux CW. Changes in Glucose Metabolism and Glycemic Status With Once-Weekly Subcutaneous Semaglutide 2.4 mg Among Participants With Prediabetes in the STEP Program. Diabetes Care. 2022 Oct 1;45(10):2396-2405. doi: 10.2337/dc21-1785. PMID 35724304
- [Derived] Wilding JPH, Batterham RL, Davies M, Van Gaal LF, Kandler K, Konakli K, Lingvay I, McGowan BM, Oral TK, Rosenstock J, Wadden TA, Wharton S, Yokote K, Kushner RF; STEP 1 Study Group. Weight regain and cardiometabolic effects after withdrawal of semaglutide: The STEP 1 trial extension. Diabetes Obes Metab. 2022 Aug;24(8):1553-1564. doi: 10.1111/dom.14725. Epub 2022 May 19. PMID 35441470
- [Derived] O'Neil PM, Birkenfeld AL, McGowan B, Mosenzon O, Pedersen SD, Wharton S, Carson CG, Jepsen CH, Kabisch M, Wilding JPH. Efficacy and safety of semaglutide compared with liraglutide and placebo for weight loss in patients with obesity: a randomised, double-blind, placebo and active controlled, dose-ranging, phase 2 trial. Lancet. 2018 Aug 25;392(10148):637-649. doi: 10.1016/S0140-6736(18)31773-2. Epub 2018 Aug 16. PMID 30122305

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 129 sites in 16 countries as follows (all sites screened and randomized): Argentina (5 sites), Belgium (5 sites), Bulgaria (5 sites), Canada (7 sites), Denmark (1 site), Finland (2 sites), France (7 sites), Germany (13 sites), India (13 sites), Japan (5 sites), Mexico (3 sites), Poland (4 sites), Russian Federation (8 sites), Taiwan(1 site), UK (10 sites), US (40 sites).
Pre-assignment Details: The trial included an initial 16-week dose-escalation period and a 52-week dose maintenance period. Participants were randomized in 2:1 ratio either to receive semaglutide 2.4 mg or placebo. The treatment is an adjunct to reduced-calorie diet and increased physical activity.
Groups:
- Semaglutide 2.4 mg: Participants were to receive once-weekly subcutaneous (s.c) injection of 0.25 mg Semaglutide administered using a PDS290 pre-filled pen-injector with a 3 mL cartridge containing Semaglutide 1.0 mg/mL or 3.0 mg/mL and followed a fixed-dose escalation regimen, with dose increases every 4 weeks (to doses of 0.5, 1.0, 1.7 and 2.4 mg/week), aiming at reaching the maintenance dose of 2.4 mg after 16 weeks. Treatment was continued on the maintenance dose of 2.4 mg Semaglutide once weekly for an additional 52 weeks until week 68. The treatment was an adjunct to a reduced-calorie diet and increased physical activity.
- Placebo: Participants were to receive once-weekly subcutaneous (s.c) injection of 0.25 mg Semaglutide placebo administered using a PDS290 pre-filled pen-injector with a 3 mL cartridge containing Semaglutide placebo 1.0 mg/mL or 3.0 mg/mL and followed a fixed-dose escalation regimen, with dose increases every 4 weeks (to doses of 0.5, 1.0, 1.7 and 2.4 mg/week), aiming at reaching the maintenance dose of 2.4 mg Semaglutide placebo after 16 weeks. Treatment was continued on the maintenance dose of 2.4 mg once weekly for an additional 52 weeks until week 68. The treatment was an adjunct to a reduced-calorie diet and increased physical activity.
Period: Overall Study
Arm/Group | Semaglutide 2.4 mg | Placebo
Started | 1306 | 655
Full Analysis Set (FAS) | 1306 | 655
Safety Analysis Set (SAS) | 1306 | 655
Completed | 1240 | 609
Not Completed | 66 | 46
Not completed — Withdrawal by Subject | 26 | 17
Not completed — Lost to Follow-up | 39 | 28
Not completed — Death | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Semaglutide 2.4 mg | Placebo | Total
Number analyzed (Participants) | 1306 | 655 | 1961
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46 (13) | 47 (12) | 46 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 955 | 498 | 1453
  Male | 351 | 157 | 508
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 150 | 86 | 236
  Not Hispanic or Latino | 1118 | 551 | 1669
  Unknown or Not Reported | 38 | 18 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 17 | 10 | 27
  Asian | 181 | 80 | 261
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 72 | 39 | 111
  White | 973 | 499 | 1472
  More than one race | 25 | 8 | 33
  Unknown or Not Reported | 38 | 17 | 55

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight (%)
Description: Change in body weight from baseline (week 0) to week 68 is presented. The endpoint was evaluated based on the data from both in-trial and on-treatment observation periods. In-trial observation period: the uninterrupted time interval from date of randomization (week 0) to date of last contact with trial site (week 75). On-treatment observation period: includes all time intervals in which participants are considered to be on treatment from the first (week 0) to last trial product administration (week 68), including 2 weeks of follow-up. It excludes any period of temporary treatment interruption. Temporary treatment interruption is defined as more than 2 consecutive missed doses (off-treatment period).
Time Frame: Baseline (week 0) to week 68
Population: Overall number of participants analyzed = full analysis set (FAS) which comprised all randomized participants. Number Analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage point
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 1306 | 655
Percentage point
  In-trial observation period: number analyzed (Participants) | 1212 | 577
  In-trial observation period | -15.6 (10.1) | -2.8 (6.5)
  On-treatment observation period: number analyzed (Participants) | 1059 | 499
  On-treatment observation period | -16.9 (9.4) | -3.1 (6.4)
Statistical Analysis 1: Comparison: Semaglutide 2.4 mg vs Placebo; Treatment policy estimand; Test type: Superiority; p < .0001, ANCOVA; Treatment difference = -12.44, 95% CI 2-sided [-13.37 to -11.51]
Statistical Analysis 2: Comparison: Semaglutide 2.4 mg vs Placebo; Hypothetical estimand; Test type: Superiority; p < 0.0001, ANCOVA; Treatment difference = -14.42, 95% CI 2-sided [-15.29 to -13.55]

2. Primary Outcome: Participants Who Achieve 5 or More Percent Body Weight Reduction (Yes/no)
Description: Number of participants who achieved weight loss more than or equal to 5% (yes/no) at week 68 are presented. The endpoint was evaluated based on the data from both in-trial and on-treatment observation periods. In-trial observation period: the uninterrupted time interval from start of randomization (week 0) to last trial-related subject-site contact (week 75). On-treatment observation period: includes all time intervals in which participants are considered to be on treatment from the first (week 0) to last trial product administration (week 68), including 2 weeks of follow-up. It excludes any period of temporary treatment interruption.
Time Frame: After week 68
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 1306 | 655
Participants
  In-trial observation period: number analyzed (Participants) | 1212 | 577
  In-trial observation period: Yes | 1047 | 182
  In-trial observation period: No | 165 | 395
  On-treatment observation period: number analyzed (Participants) | 1059 | 499
  On-treatment observation period: Yes | 978 | 165
  On-treatment observation period: No | 81 | 334
Statistical Analysis 1: Comparison: Semaglutide 2.4 mg vs Placebo; Treatment policy estimand; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 11.22, 95% CI 2-sided [8.88 to 14.19]
Statistical Analysis 2: Comparison: Semaglutide 2.4 mg vs Placebo; Hypothetical estimand; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 37.03, 95% CI 2-sided [28.02 to 48.95]

3. Secondary Outcome: Subjects Who Achieve 10 or More Percent Body Weight Reduction (Yes/no)
Description: Number of participants who achieved weight loss more than or equal to (≥) 10% at week 68 is presented. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from date of randomization (week 0) to date of last contact with trial site (week 75).
Time Frame: Week 68
Population: FAS included all randomized participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 1212 | 577
Participants
  Yes | 838 | 69
  No | 374 | 508

4. Secondary Outcome: Participants Who Achieve 15 or More Percent Body Weight Reduction (Yes/no)
Description: Number of participants who achieved more than or equal to (≥) 15% weight loss at week 68 is presented. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomization (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 1212 | 577
Participants
  Yes | 612 | 28
  No | 600 | 549

5. Secondary Outcome: Participants Who Achieve 20 or More Percent Body Weight Reduction (Yes/no)
Description: Number of participants who achieved more than or equal to (≥) 20% weight loss at week 68 is presented. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomization (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 1212 | 577
Participants
  Yes | 388 | 10
  No | 824 | 567

6. Secondary Outcome: Change in Waist Circumference (cm)
Description: Change in waist circumference from baseline (week 0) to week 68 is presented. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomization (week 0) to date of last contact with trial site (week 75).
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: Centimeter (cm)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 1210 | 575
Centimeter (cm) | -14.1 (9.6) | -4.4 (6.9)

7. Secondary Outcome: Change in Systolic Blood Pressure (mmHg)
Description: Change in systolic blood pressure from baseline (week 0) to week 68 is presented. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomization (week 0) to date of last contact with trial site (week 75).
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 1210 | 574
Millimeters of mercury (mmHg) | -7 (14) | -1 (13)

8. Secondary Outcome: Change in Short Form 36 (SF-36)
Description: SF-36 is a 36-item patient-reported survey of patient health that measures the participant's overall health-related quality of life (HRQoL). SF-36v2™ questionnaire measured eight domains of functional health and well-being as well as two component summary scores (physical component summary and mental component summary). In the metric of norm-based scores, 50 and 10 corresponds to the mean and standard deviation, respectively, for the 2009 US general population. Change from week 0 in the domain scores and component summary scores were evaluated at week 68. A positive change score indicates an improvement since baseline. These endpoints were evaluated based on the data from in-trial observation period which is the uninterrupted time interval from start of randomization (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 1195 | 566
Score on a scale
  Change in physical functioning score (SF-36) | 2.3 (6.6) | 0.4 (7.4)
  Change in SF-36 (role-physical score) | 1.1 (7.2) | -0.2 (7.2)
  Change in SF-36 (bodily pain score) | 0.5 (8.2) | -1.3 (8.9)
  Change in SF-36 (general health score) | 2.0 (7.2) | -0.6 (7.1)
  Change in SF-36 (vitality score) | 0.7 (8.0) | -1.3 (7.9)
  Change in SF-36 (social functioning score) | -0.3 (6.6) | -1.4 (7.4)
  Change in SF-36 (role-emotional score) | -0.9 (7.3) | -1.5 (7.6)
  Change in SF-36 (mental health score) | -0.8 (7.0) | -1.7 (7.4)
  Change in SF-36 (physical component summary) | 2.4 (6.7) | 0.2 (7.1)
  Change in SF-36 (mental component summary) | -1.5 (7.1) | -2.1 (7.7)

9. Secondary Outcome: Change in Impact of Weight on Quality of Life-Lite for Clinical Trial (IWQoL-Lite for CT) Score
Description: IWQoL-Lite for CT is a modified version of an instrument designed to assess weight-related quality of life. It is used to assess the impact of body weight changes on patients' physical and psychosocial functioning in three composite scores (physical function, physical and psychosocial) and a total score. The scores range between 0-100 where higher scores indicate a better quality of life. A positive change score indicates an improvement since baseline. These endpoints were evaluated based on the data from in-trial observation period which is the uninterrupted time interval from start of randomization (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomized participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 1193 | 566
Score on a scale
  Change in physical function domain score | 15.0 (21.6) | 6.0 (21.1)
  Change in physical domain score | 14.0 (20.0) | 5.0 (19.5)
  Change in psychosocial domain score | 17.4 (19.2) | 6.9 (17.8)
  Change in total score | 16.2 (17.8) | 6.3 (16.8)

10. Secondary Outcome: Change in Body Weight (kg)
Description: Change in body weight from baseline (week 0) to week 68 is presented. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomization (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomized participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: Kilogram (kg)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 1212 | 577
Kilogram (kg) | -16.1 (10.6) | -2.9 (7.2)

11. Secondary Outcome: Change in Body Mass Index (BMI) (kg/m2)
Description: Change in body mass index from baseline (week 0) to week 68 is presented. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomization (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0) to week 68
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Kilogram per square meter (kg/sqm)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 1212 | 577
Kilogram per square meter (kg/sqm) | -5.8 (3.8) | -1.0 (2.5)

12. Secondary Outcome: Change in HbA1C (%)
Description: Change in glycosylated haemoglobin (HbA1c) from baseline (week 0) to week 68 is presented. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomization (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomized participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage point of HbA1c
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 1197 | 563
Percentage point of HbA1c | -0.5 (0.3) | -0.2 (0.3)

13. Secondary Outcome: Change in HbA1C (mmol/Mol)
Description: Change in HbA1c from baseline (week 0) to week 68 is presented. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomization (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomized participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: millimoles per mole (mmol/mol)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 1197 | 563
millimoles per mole (mmol/mol) | -5.1 (3.3) | -1.8 (3.0)

14. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) (mg/dL)
Description: Change in fasting plasma glucose from baseline (week 0) to week 68 is presented. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomization (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomized participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 1175 | 557
milligrams per deciliter (mg/dL) | -9.2 (10.9) | -0.4 (12.7)

15. Secondary Outcome: Change in Fasting Serum Insulin (mIU/L) - Ratio to Baseline
Description: Change in fasting serum insulin from week 0 to week 68 is presented as ratio to baseline. Fasting serum insulin was measured in milli-international units per milliliter (mIU/mL). The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomization (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting serum insulin
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 1147 | 550
Ratio of fasting serum insulin | 0.73 (62.3) | 0.92 (56.5)

16. Secondary Outcome: Change in Diastolic Blood Pressure (mmHg)
Description: Change in diastolic blood pressure from baseline (week 0) to week 68 is presented. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomization (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomized participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 1210 | 574
Millimeters of mercury (mmHg) | -3 (9) | -1 (9)

17. Secondary Outcome: Change in Total Cholesterol (mg/dL) - Ratio to Baseline
Description: Change in fasting total cholesterol from baseline (week 0) to week 68 is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomization (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of total cholesterol
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 1196 | 561
Ratio of total cholesterol | 0.96 (14.8) | 1.00 (15.5)

18. Secondary Outcome: Change in High-density Lipoproteins (HDL) (mg/dL) - Ratio to Baseline
Description: Change in fasting HDL from baseline (week 0) to week 68 is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomization (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of HDL cholesterol
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 1192 | 558
Ratio of HDL cholesterol | 1.05 (16.1) | 1.02 (14.9)

19. Secondary Outcome: Change in Low-density Lipoproteins (LDL) (mg/dL) - Ratio to Baseline
Description: Change in fasting LDL from baseline (week 0) to week 68 is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomization (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of LDL cholesterol
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 1194 | 561
Ratio of LDL cholesterol | 0.97 (23.7) | 1.01 (25.5)

20. Secondary Outcome: Change in Very Low-density Lipoproteins (VLDL) (mg/dL) - Ratio to Baseline
Description: Change in fasting VLDL from baseline (week 0) to week 68 is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomization (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of VLDL cholesterol
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 1193 | 561
Ratio of VLDL cholesterol | 0.77 (37.7) | 0.92 (35.2)

21. Secondary Outcome: Change in Free Fatty Acids (mg/dL) - Ratio to Baseline
Description: Change in fasting free fatty acids from baseline (week 0) to week 68 is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomization (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of free fatty acids
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 1154 | 552
Ratio of free fatty acids | 0.83 (78.3) | 0.93 (70.8)

22. Secondary Outcome: Change in Triglycerides (mg/dL) - Ratio to Baseline
Description: Change in fasting triglycerides from baseline (week 0) to week 68 is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomization (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of triglycerides
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 1194 | 561
Ratio of triglycerides | 0.77 (38.3) | 0.92 (36.2)

23. Secondary Outcome: Change in High Sensitivity C-Reactive Protein (hsCRP) - (mg/L) - Ratio to Baseline
Description: Change in high sensitivity C-reactive protein from baseline (week 0) to week 68 is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomization (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of hsCRP
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 1200 | 562
Ratio of hsCRP | 0.45 (128.2) | 0.84 (102.5)

24. Secondary Outcome: Change in Plasminogen Activator Inhibitor-1 (PAI-1) Activity (AU/ml) - Ratio to Baseline
Description: Change in plasminogen activator inhibitor-1 activity from baseline (week 0) to week 68 is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomization (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of PAI-1
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 1131 | 546
Ratio of PAI-1 | 1.15 (86.5) | 1.53 (77.3)

25. Secondary Outcome: Change in Soluble Leptin Receptor (ng/mL) - Ratio to Baseline
Description: Change in soluble leptin receptor from baseline (week 0) to week 68 is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomization (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of soluble leptin receptor
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 1194 | 562
Ratio of soluble leptin receptor | 1.07 (24.9) | 1.02 (22.2)

26. Secondary Outcome: Change in Leptin (ng/mL) - Ratio to Baseline
Description: Change in leptin from baseline (week 0) to week 68 is presented as ratio to baseline. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomization (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0) to week 68
Population: FAS included all randomised participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of leptin
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 1197 | 563
Ratio of leptin | 0.52 (75.9) | 0.87 (52.7)

27. Secondary Outcome: Change in Body Composition (Total Fat Mass) (%)
Description: Change in body composition (total fat mass) from baseline (week 0) to week 68 is presented. Body composition was assessed using Dual Energy X-ray Absorpmetry (DEXA). The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomization (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0) to week 68
Population: DEXA analysis set (DXA) includes participants in the sub-population of FAS that have had a DEXA scan performed at baseline. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage point
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 83 | 39
Percentage point | -3.9 (5.4) | -0.3 (2.8)

28. Secondary Outcome: Change in Body Composition (Total Fat Mass) (kg)
Description: as for outcome 27
Time Frame: Baseline (week 0) to week 68
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 83 | 39
Kilograms | -9.3 (8.5) | -1.5 (5.1)

29. Secondary Outcome: Change in Body Composition (Lean Body Mass) (%)
Description: Change in body composition (lean body mass) from baseline (week 0) to week 68 is presented. Body composition was assessed using DEXA. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomization (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0) to week 68
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Percentage point
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 83 | 39
Percentage point | 3.4 (5.1) | 0.2 (2.7)

30. Secondary Outcome: Change in Body Composition (Lean Body Mass) (kg)
Description: as for outcome 29
Time Frame: Baseline (week 0) to week 68
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 83 | 39
Kilograms | -5.8 (4.6) | -1.8 (2.5)

31. Secondary Outcome: Change in Body Composition (Visceral Fat Mass) (%)
Description: Change in body composition (visceral fat mass) from baseline (week 0) to week 68 is presented. Body composition was assessed using DEXA. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomization (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0) to week 68
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Percentage point
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 83 | 39
Percentage point | -2.2 (4.4) | -0.1 (4.5)

32. Secondary Outcome: Change in Body Composition (Visceral Fat Mass) (kg)
Description: as for outcome 31
Time Frame: Baseline (week 0) to week 68
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 83 | 39
Kilograms | -0.4 (0.3) | -0.1 (0.3)

33. Secondary Outcome: Change in Body Weight (%) - DEXA Subpopulation
Description: Change in body weight from baseline (week 0) to week 68 is presented in DEXA subpopulation. The endpoint was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomization (week 0) to last trial-related subject-site contact (week 75).
Time Frame: Baseline (week 0) to week 68
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Percentage point
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 89 | 42
Percentage point | -15.8 (11.1) | -3.4 (6.1)

34. Secondary Outcome: Change in Body Weight (kg) - DEXA Subpopulation
Description: as for outcome 33
Time Frame: Baseline (week 0) to week 68
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 89 | 42
Kilograms | -15.5 (11.4) | -3.2 (6.1)

35. Secondary Outcome: Participants Who Achieve "Responder Definition Value" (Yes/no) for SF-36 Physical Functioning Score
Description: The observed number of participants experiencing a meaningful within participant improvement in SF-36 Physical function after 68 weeks was determined based on two different thresholds. The threshold of 4.3 is the default generic responder threshold defined in SF-36 manual for a general population. The threshold of 3.7 is specific for the population with overweight or obesity included in the study and calculated using patient global rating anchor questionnaires to reflect participants' own perspective based on FDA recommendations. In the reported data, "Yes" infers the number of participants who have achieved an improvement in score greater than or equal to the threshold and "No" infers number of participants who have not achieved an improvement in score greater than or equal to the threshold. The endpoint was evaluated based on the in-trial observation period which is the uninterrupted time interval from randomization (week 0) to last trial related subject-site contact (week 75).
Time Frame: After week 68
Population: FAS included all randomized participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 1195 | 566
Participants
  Yes (with threshold 4.3) | 318 | 97
  No (with threshold 4.3) | 877 | 469
  Yes (with threshold 3.7) | 478 | 153
  No (with threshold 3.7) | 717 | 413

36. Secondary Outcome: Participants Who Achieve "Responder Definition Value" (Yes/no) for IWQoL-Lite for CT Physical Function Domain (5-items) Score
Description: The observed number of participants experiencing a meaningful within participant improvement in IWQOL-Lite-CT physical function after 68 weeks was determined based on two different thresholds. The threshold of 20 was a preliminary responder threshold based on earlier studies. The threshold of 14.6 is specific for the population with overweight or obesity included in the study and calculated using patient global rating anchor questionnaires to reflect participants' own perspective based on FDA recommendations. In the reported data, "Yes" infers the number of participants who have achieved an improvement in score greater than or equal to the threshold and "No" infers the number of participants who have not achieved an improvement in score greater than or equal to the threshold. The endpoint was evaluated based on the in-trial observation period. In trial observation period: the uninterrupted time interval from randomization (week 0) to last trial related subject-site contact (week 75).
Time Frame: After week 68
Population: FAS included all randomized participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 1193 | 566
Participants
  Yes (with threshold 20) | 473 | 145
  No (with threshold 20) | 720 | 421
  Yes (with threshold 14.6) | 611 | 186
  No (with threshold 14.6) | 582 | 380

37. Secondary Outcome: Number of Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a product, whether or not considered related to the product. All AEs mentioned here are treatment emergent adverse events (TEAE) defined as an event for which the onset of the event occurs in the on-treatment period. The endpoint was evaluated based on the data from on-treatment observation period. On-treatment observation period: includes all time intervals in which participants are considered to be on treatment from the first (week 0) to last trial product administration (week 68), including 7 weeks of follow-up. It excludes any period of temporary treatment interruption. Temporary treatment interruption is defined as more than 7 consecutive missed doses (off-treatment period).
Time Frame: Baseline (week 0) to week 75
Population: SAS included all participants who received at least one dose of trial product.
Measure: Number; unit: Events
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 1306 | 655
Events | 9658 | 3302

38. Secondary Outcome: Number of Serious Adverse Events (SAEs)
Description: A serious adverse event (SAE) is defined as any untoward medical occurrence that at any dose results in death, or is life-threatening, or requires inpatient hospitalization or causes prolongation of existing hospitalization results in persistent or significant disability/incapacity, or may have caused a congenital anomaly/birth defect, or requires intervention to prevent permanent impairment or damage. The SAEs occurred from week 0 to week 75 is presented. The endpoint was evaluated based on the data from on-treatment observation period. On-treatment observation period: includes all time intervals in which participants are considered to be on treatment from the first (week 0) to last trial product administration (week 68), including 7 weeks of follow-up. It excludes any period of temporary treatment interruption. Temporary treatment interruption is defined as more than 7 consecutive missed doses (off-treatment period).
Time Frame: Baseline (week 0) to week 75
Population: SAS included all participants who received at least one dose of trial product.
Measure: Number; unit: Events
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 1306 | 655
Events | 164 | 53

39. Secondary Outcome: Change in Pulse
Description: Change in pulse from baseline (week 0) to week 68 is presented. The endpoint was evaluated based on the data from on-treatment observation period. On-treatment observation period: includes all time intervals in which participants are considered to be on treatment from the first (week 0) to last trial product administration (week 68) including 2 weeks of follow-up. It excludes any period of temporary treatment interruption. Temporary treatment interruption is defined as more than 2 consecutive missed doses (off-treatment period).
Time Frame: Baseline (week 0) to week 68
Population: SAS included all participants who received at least one dose of trial product. Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 1059 | 499
beats per minute (bpm) | 3 (10) | -1 (10)

40. Secondary Outcome: Change in Amylase - Ratio to Baseline
Description: Change in amylase (measured as units per litre [U/L]) is presented as ratio to baseline. The endpoint was evaluated based on the data from on-treatment observation period. On-treatment observation period: includes all time intervals in which participants are considered to be on treatment from the first (week 0) to last trial product administration (week 68) including 2 weeks of follow-up. It excludes any period of temporary treatment interruption. Temporary treatment interruption is defined as more than 2 consecutive missed doses (off-treatment period).
Time Frame: Baseline (week 0) to week 68
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of amylase
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 1053 | 497
Ratio of amylase | 1.14 (21.6) | 1.03 (21.4)

41. Secondary Outcome: Change in Lipase - Ratio to Baseline
Description: Change in lipase (measured as units per litre [U/L]) is presented as ratio to baseline. The endpoint was evaluated based on the data from on-treatment observation period. On-treatment observation period: includes all time intervals in which participants are considered to be on treatment from the first (week 0) to last trial product administration (week 68) including 2 weeks of follow-up. It excludes any period of temporary treatment interruption. Temporary treatment interruption is defined as more than 2 consecutive missed doses (off-treatment period).
Time Frame: Baseline (week 0) to week 68
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of lipase
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 1053 | 496
Ratio of lipase | 1.41 (49.3) | 0.97 (37.3)

42. Secondary Outcome: Change in Calcitonin - Ratio to Baseline
Description: Change in calcitonin (measured as ng/L) is presented as ratio to baseline. The endpoint was evaluated based on the data from on-treatment observation period. On-treatment observation period: includes all time intervals in which participants are considered to be on treatment from the first (week 0) to last trial product administration (week 68) including 2 weeks of follow-up. It excludes any period of temporary treatment interruption. Temporary treatment interruption is defined as more than 2 consecutive missed doses (off-treatment period).
Time Frame: Baseline (week 0) to week 68
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of calcitonin
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 1050 | 497
Ratio of calcitonin | 0.99 (37.6) | 0.95 (40.9)

ADVERSE EVENTS:
Time Frame: week 0 to week 75 Results are based on the SAS which included all participants who received at least one dose of Semaglutide or placebo.
Description: All AEs mentioned here are TEAE defined as an event that had onset date (or increase in severity) on or after the first day of exposure to randomized treatment and no later than the date of last dose + 7 weeks.
Groups:
- Sema 2.4 mg: Participants were to receive once-weekly subcutaneous (s.c) injection of 0.25 mg Semaglutide administered using a PDS290 pre-filled pen-injector with a 3 mL cartridge containing Semaglutide 1.0 mg/mL or 3.0 mg/mL and followed a fixed-dose escalation regimen, with dose increases every 4 weeks (to doses of 0.5, 1.0, 1.7 and 2.4 mg/week), aiming at reaching the maintenance dose of 2.4 mg after 16 weeks. Treatment was continued on the maintenance dose of 2.4 mg Semaglutide once weekly for an additional 52 weeks until week 68. The treatment was an adjunct to a reduced-calorie diet and increased physical activity.
Arm/Group | Sema 2.4 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 1/1306 | 1/655
Serious Adverse Events (participants affected / at risk) | 128/1306 | 42/655
Other Adverse Events (participants affected / at risk) | 1052/1306 | 447/655
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sema 2.4 mg (N=1306) | Placebo (N=655)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominoplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Acute stress disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 5 (5) | 1 (1)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0)
Arthritis infective (Infections and infestations) | 0 (0) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 2 (4) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bacterial colitis (Infections and infestations) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bone prosthesis insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 4 (4) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 3 (3) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 12 (12) | 1 (1)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cranial nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Gastric bypass (Surgical and medical procedures) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 5 (5) | 0 (0)
Gastroenteritis astroviral (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hairy cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hepatitis E (Infections and infestations) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hip surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Idiopathic intracranial hypertension (Nervous system disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Large intestine infection (Infections and infestations) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Meningitis viral (Infections and infestations) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nerve compression (Nervous system disorders) | 1 (1) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0)
Oesophageal achalasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Optic ischaemic neuropathy (Eye disorders) | 2 (2) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Psychogenic seizure (Nervous system disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pyelonephritis (Infections and infestations) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Splenic haemorrhage (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Toxoplasmosis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Uterine haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vascular stent occlusion (General disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 0 (0)
Vertigo CNS origin (Nervous system disorders) | 1 (1) | 0 (0)
Volvulus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 0 (0)
Weight increased (Investigations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sema 2.4 mg (N=1306) | Placebo (N=655)
Abdominal distension (Gastrointestinal disorders) | 96 (135) | 31 (42)
Abdominal pain (Gastrointestinal disorders) | 127 (172) | 36 (41)
Abdominal pain upper (Gastrointestinal disorders) | 125 (176) | 35 (37)
Arthralgia (Musculoskeletal and connective tissue disorders) | 81 (92) | 43 (47)
Back pain (Musculoskeletal and connective tissue disorders) | 106 (120) | 53 (55)
Constipation (Gastrointestinal disorders) | 305 (389) | 62 (73)
Cough (Respiratory, thoracic and mediastinal disorders) | 40 (45) | 33 (35)
Decreased appetite (Metabolism and nutrition disorders) | 124 (139) | 22 (26)
Diarrhoea (Gastrointestinal disorders) | 411 (765) | 104 (138)
Dizziness (Nervous system disorders) | 98 (129) | 23 (35)
Dyspepsia (Gastrointestinal disorders) | 135 (179) | 23 (30)
Eructation (Gastrointestinal disorders) | 112 (139) | 3 (3)
Fatigue (General disorders) | 104 (120) | 28 (29)
Gastroenteritis (Infections and infestations) | 81 (99) | 30 (38)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 82 (92) | 20 (21)
Headache (Nervous system disorders) | 198 (386) | 80 (104)
Influenza (Infections and infestations) | 89 (112) | 63 (79)
Nasopharyngitis (Infections and infestations) | 281 (480) | 133 (216)
Nausea (Gastrointestinal disorders) | 576 (1067) | 114 (146)
Sinusitis (Infections and infestations) | 70 (83) | 36 (40)
Upper respiratory tract infection (Infections and infestations) | 114 (158) | 80 (116)
Urinary tract infection (Infections and infestations) | 68 (83) | 28 (33)
Vomiting (Gastrointestinal disorders) | 321 (632) | 43 (52)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property

DOCUMENTS (2):
  • Study Protocol (2019-03-29): https://cdn.clinicaltrials.gov/large-docs/35/NCT03548935/Prot_002.pdf
  • Statistical Analysis Plan (2020-07-03): https://cdn.clinicaltrials.gov/large-docs/35/NCT03548935/SAP_003.pdf